CLINICAL TRIAL: NCT00536029
Title: MicroRNA Expression and Function in Cutaneous Malignant Melanoma
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: H-C-2007-0009
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2007-09

CONDITIONS: Melanoma
Keywords: Melanoma; SIAscope; pigmented skin lesions
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Subject with pigmented skin lesion suspect for malignant melanoma

SUMMARY:
Spectrophotometric intracutaneous analysis (SIAscopy) is a new technique for imaging pigmented skin lesions and for diagnosing melanoma and non-melanoma skin cancer. The SIAscope is a portable system comprising of a laptop computer connected to a small handheld skin probe equipped with a light source. The skin lesion is interrogated with light of different wavelengths and the reflection spectra analysed by proprietary algorithms showing distribution, position and quantity of melanin, blood and collagen within the papillary dermis (the SIAgraphs). Earlier studies generated promising results and documented >80% specificity and sensitivity of SIAscopy for melanoma diagnosis. It has been suggested that this technique could be used for the initial screening and selection of pigmented lesion for excision. In this work we addressed the usefulness of SIAscopy for the clinical diagnosis of pigmented malignant melanoma in a prospective, blinded design.

ELIGIBILITY:
Inclusion Criteria:

* Pigmented lesion

Exclusion Criteria:

* No pigmented lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-02; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Glud, Cand.med., Principal Investigator — Department for Plastic Surgery and Burn Unit
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Govindan K, Smith J, Knowles L, Harvey A, Townsend P, Kenealy J. Assessment of nurse-led screening of pigmented lesions using SIAscope. J Plast Reconstr Aesthet Surg. 2007;60(6):639-45. doi: 10.1016/j.bjps.2006.10.003. Epub 2007 Jan 31. PMID 17485052
- [Background] Haniffa MA, Lloyd JJ, Lawrence CM. The use of a spectrophotometric intracutaneous analysis device in the real-time diagnosis of melanoma in the setting of a melanoma screening clinic. Br J Dermatol. 2007 Jun;156(6):1350-2. doi: 10.1111/j.1365-2133.2007.07932.x. PMID 17535234
- [Background] Moncrieff M, Cotton S, Claridge E, Hall P. Spectrophotometric intracutaneous analysis: a new technique for imaging pigmented skin lesions. Br J Dermatol. 2002 Mar;146(3):448-57. doi: 10.1046/j.1365-2133.2002.04569.x. PMID 11952545